CLINICAL TRIAL: NCT04552119
Title: Prospective, Multi-Center, Post-Market Clinical Follow-up Study to Evaluate Safety and Performance of the HEALICOIL™ Knotless Suture Anchor in Shoulder Rotator Cuff Tendon Repair
Brief Title: Safety of Treatment of Shoulder Repair
Acronym: HEALICOIL_KNTL
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HEALICOIL.KNOTLESS.2019.12
Record Dates: First submitted 2020-09-09; First posted 2020-09-17 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Rotator Cuff
Keywords: Rotator cuff; shoulder repair; HEALICOIL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HEALICOIL Knotless Suture REGENESORB: HEALICOIL™ Knotless Suture Anchor in Shoulder Rotator Cuff Tendon Repair using HEALICOIL Knotless REGENESORB
  Interventions: Device: HEALICOIL Knotless REGENESORB
- HEALICOIL Knotless PEEK: HEALICOIL™ Knotless Suture Anchor in Shoulder Rotator Cuff Tendon Repair using HEALICOIL Knotless PEEK
  Interventions: Device: HEALICOIL Knotless PEEK

INTERVENTIONS:
Device: HEALICOIL Knotless PEEK — HEALICOIL Knotless PEEK Self-Tapping HEALICOIL Knotless Non-Self Tapping
  Groups: HEALICOIL Knotless PEEK
Device: HEALICOIL Knotless REGENESORB — HEALICOIL Knotless REGENESORB Self -Tapping HEALICOIL Knotless REGENSORB Non-Self Tapping
  Groups: HEALICOIL Knotless Suture REGENESORB

SUMMARY:
This study evaluates the safety of the HEALICOIL Knotless Suture Anchors in patients requiring a repair of the rotator cuff tendon repair

DETAILED DESCRIPTION:
This is a multicenter, prospective, post-marketing, observational, case series study to evaluate the safety and efficacy of the HEALICOIL Knotless Suture Anchors in subjects with rotator cuff tendon repair. Approximately 160 subjects will be enrolled at up to 6 sites. Safety monitoring will include documentation device- and surgery-related AEs. Efficacy will be monitored by assessment of post-operative follow up, clinical complications, reoperation rate, EQ-5D-5L, and pain VAS.

ELIGIBILITY:
Inclusion Criteria:

1. Requires reattachment of soft tissue to bone for the following shoulder indications:

   1. Rotator Cuff Tendon repair

      * i. Single or double row rotator cuff repair using HEALICOIL Knotless PEEK NST, HEALICOIL Knotless PEEK Self-Tapping, or HEALICOIL Knotless RG Self-Tapping; OR
      * ii. Double row rotator cuff repair using HEALICOIL Knotless RG NST in lateral row (existing HEALICOIL RG device to be used in medial row of the repair); AND/OR
   2. Biceps tenodesis

      * i. In conjunction with Rotator Cuff Tendon repair using HEALICOIL Knotless PEEK NST, HEALICOIL Knotless PEEK Self-Tapping, HEALICOIL Knotless RG NST or HEALICOIL Knotless RG Self-Tapping OR
      * ii. As a stand-alone procedure for HEALICOIL Knotless PEEK NST, HEALICOIL Knotless PEEK Self-Tapping, or HEALICOIL Knotless RG Self-Tapping (not HEALICOIL Knotless RG NST
2. Has a pre-operative standard of care MRI within 6 months of surgery containing the following sequences:

   1. Sat T2 FS: Oblique Sag T2-weighted Fat Saturation Spin Echo (oriented perpendicular to the scapula), with TE > 70 ms, AND
   2. Cor T2 FS: Oblique Cor T2-weighted Fat Saturation Spin Echo (oriented parallel to the scapula), with TE > 70 ms, AND
   3. Sag T1: Oblique Sag T1-weighted Spin Echo (oriented perpendicular to the scapula); OR
   4. Willing and able to undergo an additional study specific pre-operative MRI according to the study Imaging Protocol if the above criteria is not met OR
   5. MRI not required; subject not in HEALICOIL RG NST subgroup
3. Has consented to participate in the study by signing the IRB/IEC approved informed consent form.
4. Requires only one variant of the HEALICOIL Knotless Suture Anchor
5. Is ≥18 years of age at time of surgery
6. Willing and able to make all required study visits
7. Able to follow instructions (Approved translated documents supplied upon request)

Exclusion Criteria:

* Any one (1) of the following criteria will disqualify a potential subject from participation in the study:

  1. Known hypersensitivity to the implant material. Where material sensitivity is suspected, appropriate tests should be made and sensitivity ruled out prior to implantation.
  2. Pathological conditions of bone, such as cystic changes or severe osteopenia, which would compromise secure anchor fixation.
  3. Pathological conditions in the soft tissues to be attached that would impair secure fixation by suture.
  4. Comminuted bone surface, which would compromise secure anchor fixation.
  5. Physical conditions which would eliminate, or tend to eliminate, adequate anchor support or retard healing
  6. The presence of infection.
  7. Conditions which would limit the subject's ability or willingness to restrict activities or follow directions during the healing period.
  8. Concurrent bilateral surgery.
  9. Participation in the treatment period of another clinical trial within thirty (30) days of Visit 1, or during the study.
  10. Women who are pregnant.
  11. Prior ipsilateral surgeries performed on the joint space.
  12. Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Repair failure rate of HEALICOIL Knotless Suture Anchors | 6 months
  Repair failure rate defined as the need for a second repair procedure at 6 months.

SECONDARY OUTCOMES:
Repair failure rate at 12 months and 24 months | 12 and 24 months
  Repair failure rate is defined as the need for a second repair procedure. Repair rate at 24 months will be collected for the HEALICOIL Knotless REGENESORB Non-Self Tapping subgroup only.
Constant-Murley Score | 6, 12, and 24 months
  Constant-Murley Shoulder (CMS) scale assesses four aspects related to shoulder pathology; two subjective: pain and activities of daily living (ADL) and two objective: range of motion (ROM) and strength. The subjective components can receive up to 35 points and the objective 65, resulting in a possible maximum total score of 100 points (best function). Pain and ADL are answered by the subject; ROM and strength require a physical evaluation and are answered by the orthopaedic surgeon or the physiotherapist.
American Shoulder and Elbow Surgeons (ASES) Visual Analog Scale (VAS) pain score | 6, 12, and 24 months
  The ASES instrument is composed of 2 sections containing participant self-reported and clinician assessments. The ASES score is a 0 to 100-point rating with a higher score indicating improvement in pain and function. It is based solely on participant responses and is a combination of the participant's shoulder pain rating (VAS Pain) and self-reported ability to perform 10 different activities of daily living (ADLs).
Single Assessment Numeric Evaluation (SANE) Shoulder scale at 6 months and 12 months | 6 and 12 months
  The SANE is a simple, single-question, patient-based shoulder function assessment tool: ''How would you rate your shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?''
EQ-5D-3L at 6 months and 12 months | 6 and 12 months
  The EuroQol EQ-5D-3L is a descriptive system measuring health-related Quality Of Life (QOL) and consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which takes one of three responses. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D-3L dimension.
Tendon thickening and anchor absorption/replacement by bone at 6 months and 24 months for HEALICOIL Knotless REGENESORB Non-Self Tapping | 6 and 24 months
  Magnetic Resonance Imaging (MRI) will be used to determine tendon thickening and anchor absorption/replacement by bone at 6 and 24 months.
Tendon re-tear rate at 6 months and 24 months for HEALICOIL Knotless REGENESORB Non-Self Tapping only | 6 and 24 months
  Magnetic Resonance Imaging (MRI) will be used to determine tendon re-tear rate at 6 months and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Karlie Morgan, Study Chair — Smith & Nephew, Inc.
Locations (5):
- United States (5):
  - University of Stanford, Redwood City, California
  - Orthopaedic and Spine Center of Southern Colorado, Colorado Springs, Colorado
  - University of Colorado - Denver, Denver, Colorado
  - OrthoIllinois LTD, Rockford, Illinois
  - University Orthopedics Center, Altoona, Pennsylvania

IPD SHARING:
Plan to Share IPD: No